CLINICAL TRIAL: NCT00304889
Title: Vancomycin Vs. Nitazoxanide to Treat Clostridium Difficile Colitis That Has Failed Therapy With Metronidazole
Brief Title: Vancomycin vs. Nitazoxanide to Treat Recurrent C. Difficile Colitis
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Daniel M. Musher MD, Principle Investigator, Michael E. DeBakey VA Medical Center
Other Study IDs: H-18736
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2013-02

CONDITIONS: Clostridium Enterocolitis; Pseudomembranous Colitis; Antibiotic-Associated Colitis
Keywords: Clostridium difficile
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to compare the outcome of treatment with nitazoxanide vs. vancomycin for diarrheal disease due to Clostridium difficile in patients who have failed previous treatment with metronidazole.

DETAILED DESCRIPTION:
Clostridium difficile is the leading cause of nosocomial diarrheal disease associated with antibiotic therapy. This is a debilitating condition with substantial morbidity and a mortality that used to be said to be around 2-3%, but that has recently been shown by us (Clin Infect. Dis, July, 2005) and others (Pepin et al, Clin. Infect. Dis., July, 2005) to be substantially higher -- approximately 15-20%. There has been an enormous increase in this disease at the VA medical center during the past two years, just as has occurred at other hospitals throughout the United States and the developed world.

Although orally administered vancomycin was the first drug to be approved in treating C. difficile colitis, and remains the only one with the official approval by the Food and Drug Administration, the currently recommended therapy for this condition is metronidazole, given orally. This drug was recommended because: (1) the cost of vancomycin was exceedingly high; (2) there was concern that vancomycin-resistant bacteria might appear in hospitals if the drug was used to treat large number of patients; and (3) these recommendations were made at a time that the cure rate from metronidazole was thought to approach 100%.

We have recently shown that 23% of patients fail to respond to initial therapy with metronidazole, and another 27% relapse after treatment (Musher et al, Clin Infect Dis, July, 2005). Others have confirmed these observations (Pepin et al, Clin Infect Dis, July 2005). The options for treating failure or relapse are limited. Another course of metronidazole may cure about one-half of patients. Oral vancomycin may be used, but this drug also has a failure rate of 10-20% and the concerns about its use remain.

Based on this background, we became interested in studying nitazoxanide. This is an FDA approved drug, marketed in the United States and widely used throughout the world to treat parasitic diseases of the gastrointestinal tract; several million children have been treated with this drug during the past decade. The drug acts by interfering with anaerobic metabolic pathways, and it has been shown to have excellent in vitro activity against C. difficile. We hypothesized that this drug was both safe and effective as an alternative in patients who have diarrheal disease caused by C. difficile. The IRB approved a double-blind protocol to compare metronidazole with nitazoxanide, and we have completed that trial.

The results of this study were very favorable. A 10-day course of oral nitazoxanide produced a cure of symptoms at 7 days of about 90% and a cure without relapse at 31 days of about 79% compared to 84% and 56%, respectively, for metronidazole. Because of the small numbers of subjects, these differences were not statistically significant, but the results certainly appeared promising. A manuscript has just been submitted to Clin Infect Dis describing this study.

We now propose to compare nitazoxanide to vancomycin in the group of patients most in need of alternative therapy, namely those who have been treated with metronidazole and have failed or have had a recurrence of disease after an initial response.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* clinical diagnosis of C. difficile associated disease, based on the new onset of diarrhea, abdominal discomfort, or otherwise unexplained fever or leukocytosis
* diagnosis of C. difficile colitis proven by positive assay for C. difficile toxin in feces
* disease has been treated, and the symptoms failed to respond to treatment with metronidazole, or symptoms recurred after the patient has completed a course of metronidazole therapy
* able to take oral medication

Exclusion Criteria:

* patients with other recognized causes of diarrhea or colitis
* women of child bearing age who are pregnant, breast feeding, or not using birth control
* patients of known causes of diarrhea, such as inflammatory bowel disease
* patients in whom diarrhea can not be evaluated, such as those with colostomy
* patients with renal insufficiency (BUN or creatinine >3.0 times baseline)
* patients who are medically unstable, for example in an ICU and on medications to maintain blood pressure
* patients who are regarded as unlikely to survive for 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for C. difficile.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Days to symptom resolution | observation
  Number of day to resolution to three formed or loose stools per day

SECONDARY OUTCOMES:
side effects | observational
  number of side effects from medication

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Houston VA Medical Center, Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States